CLINICAL TRIAL: NCT00817713
Title: Can Anthelminthic Treatment Delay the Progression of HIV? Randomised Open-label Trial Testing Presumptive Anthelminthic Treatment on Progression of HIV in ART-naïve HIV-positive Patients in a Rural African Setting With Presumed High Prevalence of Helminth Infections.
Brief Title: Can Presumptive Anthelminthic Treatment Delay the Progression of HIV in ART-naïve Patients in Rural Africa?
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated prematurely due to recruitment difficulties. Expansion to more study sites not planned.
Sponsor: Swiss Tropical & Public Health Institute (Other)
Collaborators: Ifakara Health Research and Development Centre (Other); Insel Gruppe AG, University Hospital Bern (Other); Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Cornelia Staehelin, MD, Swiss Tropical Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 257/08
Record Dates: First submitted 2009-01-05; First posted 2009-01-06 (Estimated); Last update posted 2011-02-16 (Estimated); Status verified 2009-04

CONDITIONS: HIV Infections; Helminthiasis
Keywords: Human Immunodeficiency Virus; Helminthiasis; treatment naive; co-infection; immune modulation
MeSH Terms: conditions — HIV Infections; Helminthiasis; Acquired Immunodeficiency Syndrome; Coinfection | interventions — Praziquantel; Ivermectin; Albendazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- anthelminthic treatment (Active Comparator): Albendazol plus fix-dose Praziquantel plus Ivermectin
  Interventions: Drug: Praziquantel, Ivermectin, Albendazole
- HIV care, no anthelminthic treatment (No Intervention): HIV care as per Tanzanian National AIDS Control Program (NACP) guidelines

INTERVENTIONS:
Drug: Praziquantel, Ivermectin, Albendazole — Standard HIV care plus triple anthelminthic treatment
  * Praziquantel 2400mg single dose
  * Ivermectin 12 mg, single dose
  * Albendazole 400mg, 2 doses in 1 day
  All drugs given at baseline, after 6 months and after 12 months.
  Arms: anthelminthic treatment

SUMMARY:
This study focuses on one of the major health issues of Sub-Saharan Africa: multi-parasitism and co-infections. In particular this study aims to elucidate the interaction of helminths with HIV.

There is good reason to suspect a detrimental effect of helminth infection on the course of HIV infection. We hypothesize, that treatment of helminths in HIV- and helminth co-infected individuals leads to a reduction of HIV viral load. With a lower HIV RNA level one would expect a slower decline of CD4 cells and hence also a slower progression of the disease. Ideally this would lead to a prolongation of the chronic phase of HIV infection and to a delay in the time when anti-retroviral treatment needs to be started.

DETAILED DESCRIPTION:
* Background: On the basis of immunological considerations and in vitro trials on co-infections there is strong reason to suspect a detrimental effect of helminth infection on the course of HIV. The immunological answer very efficiently evoked by helminth infection is aimed at hijacking and suppressing the immune system in order to suit the requirements of the specific helminth. This permits helminths to cause chronic infection, often persisting over years and allowing some infecting worms to grow to several centimetres of length within their host. However, this immune modulation also affects non-related antigens (for example HIV) which would actually require a different line of immunological action.

Some clinical trials have been able to confirm this detrimental effect of helminths on HIV infection, while other trials failed to do so. A recent Cochrane review on clinical trials with HIV and helminth co-infection found an overall slight reduction of HIV viral load if helminth infection was treated. However there was no measurable effect on CD4 count or clinical staging of HIV. This might be explained by the fact that these trials were very heterogeneous in their set-up and were run for too short a time (max 6 months) to allow sufficient answers to these questions.

According to mathematical models, even a relatively modest reduction of HIV RNA by 0.5 log could delay the need to start combined antiretroviral therapy by about 3.5 years and potentially prolong the symptom-free phase of HIV-infection by nearly 1 year. On a population scale this could lead to substantial savings with regard to drug and clinical costs and on an individual level to an invaluable gain in drug-free and ideally also symptom-free life years.

* Objective: To assess the impact of presumptive anthelminthic treatment on HIV progression in patients infected with HIV in a rural setting with presumed high prevalence of helminth infection.
* Methods: Randomised open-label trial of presumptive triple anthelminthic treatment in HIV positive patients not yet requiring anti-retroviral treatment.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive patients
* most recent CD4-count > 250 c/μl (latest within the previous 7 months)
* anti-retroviral treatment naïve
* age >18 years
* provide written informed consent

Exclusion Criteria:

* Pregnant and lactating women in the first week of lactation
* Symptoms of severe anemia (or haemoglobin <5g/dl within the precious 3 months)
* Symptoms of chronic diarrhea (defined as >= 3 stools per day of loose consistency for more than 2 weeks)
* Patients on treatment for tuberculosis
* WHO clinical stage 3 disease and CD4-count <350 c/μl
* WHO clinical stage 4 disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 295 (Actual)
Dates: Start 2009-01; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Difference in HIV viral load between intervention and control arm | one year

SECONDARY OUTCOMES:
Difference in CD4 counts between intervention and control arm | one year
Difference in time to meet criteria for the initiation of anti-retroviral treatment | one year
occurrence of severe adverse events | one year

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia J. Staehelin, MD, Principal Investigator — Swiss Tropical Institute, Ifakara Health Institute; Christoph F. Hatz, MD, Prof., Study Director — Swiss Tropical & Public Health Institute; Hansjakob Furrer, MD, Prof., Study Chair — Infectious Disease Unit, Inselspital, University Hospital Berne, 3010 Berne, Switzerland; Honorathy Urassa, MSc, Study Chair — Ifakara Health Institute; Baraka Amuri, MD, Principal Investigator — Ifakara Health Institute; Salim Hamis, MD, Study Chair — Ifakara Health Institute; Juerg Utzinger, Prof., Study Chair — Swiss Tropical & Public Health Institute; Erik Mossdorf, MD, Study Chair — Swiss Tropical & Public Health Institute
Locations (1):
- Chronic Disease Clinic of St. Francis Designated District Hospital, Ifakara, Kilombero, Tanzania

REFERENCES:
- [Background] Walson JL, John-Stewart G. Treatment of helminth co-infection in HIV-1 infected individuals in resource-limited settings. Cochrane Database Syst Rev. 2008 Jan 23;(1):CD006419. doi: 10.1002/14651858.CD006419.pub2. PMID 18254104
- [Background] Walson JL, Otieno PA, Mbuchi M, Richardson BA, Lohman-Payne B, Macharia SW, Overbaugh J, Berkley J, Sanders EJ, Chung MH, John-Stewart GC. Albendazole treatment of HIV-1 and helminth co-infection: a randomized, double-blind, placebo-controlled trial. AIDS. 2008 Aug 20;22(13):1601-9. doi: 10.1097/QAD.0b013e32830a502e. PMID 18670219
- [Background] Gupta SB, Jacobson LP, Margolick JB, Rinaldo CR, Phair JP, Jamieson BD, Mehrotra DV, Robertson MN, Straus WL. Estimating the benefit of an HIV-1 vaccine that reduces viral load set point. J Infect Dis. 2007 Feb 15;195(4):546-50. doi: 10.1086/510909. Epub 2007 Jan 5. PMID 17230414
- [Background] Mohammed KA, Haji HJ, Gabrielli AF, Mubila L, Biswas G, Chitsulo L, Bradley MH, Engels D, Savioli L, Molyneux DH. Triple co-administration of ivermectin, albendazole and praziquantel in zanzibar: a safety study. PLoS Negl Trop Dis. 2008 Jan 23;2(1):e171. doi: 10.1371/journal.pntd.0000171. PMID 18235853
- [Background] Brown M, Mawa PA, Kaleebu P, Elliott AM. Helminths and HIV infection: epidemiological observations on immunological hypotheses. Parasite Immunol. 2006 Nov;28(11):613-23. doi: 10.1111/j.1365-3024.2006.00904.x. PMID 17042933
- [Background] Kallestrup P, Zinyama R, Gomo E, Butterworth AE, Mudenge B, van Dam GJ, Gerstoft J, Erikstrup C, Ullum H. Schistosomiasis and HIV-1 infection in rural Zimbabwe: effect of treatment of schistosomiasis on CD4 cell count and plasma HIV-1 RNA load. J Infect Dis. 2005 Dec 1;192(11):1956-61. doi: 10.1086/497696. Epub 2005 Oct 20. PMID 16267767
- [Background] Brown M, Kizza M, Watera C, Quigley MA, Rowland S, Hughes P, Whitworth JA, Elliott AM. Helminth infection is not associated with faster progression of HIV disease in coinfected adults in Uganda. J Infect Dis. 2004 Nov 15;190(10):1869-79. doi: 10.1086/425042. Epub 2004 Oct 20. PMID 15499545
- [Background] Elliott AM, Mawa PA, Joseph S, Namujju PB, Kizza M, Nakiyingi JS, Watera C, Dunne DW, Whitworth JA. Associations between helminth infection and CD4+ T cell count, viral load and cytokine responses in HIV-1-infected Ugandan adults. Trans R Soc Trop Med Hyg. 2003 Jan-Feb;97(1):103-8. doi: 10.1016/s0035-9203(03)90040-x. PMID 12886815
- [Background] Modjarrad K, Zulu I, Redden DT, Njobvu L, Lane HC, Bentwich Z, Vermund SH. Treatment of intestinal helminths does not reduce plasma concentrations of HIV-1 RNA in coinfected Zambian adults. J Infect Dis. 2005 Oct 1;192(7):1277-83. doi: 10.1086/444543. Epub 2005 Aug 25. PMID 16136473
- [Background] Wolday D, Mayaan S, Mariam ZG, Berhe N, Seboxa T, Britton S, Galai N, Landay A, Bentwich Z. Treatment of intestinal worms is associated with decreased HIV plasma viral load. J Acquir Immune Defic Syndr. 2002 Sep 1;31(1):56-62. doi: 10.1097/00126334-200209010-00008. PMID 12352151